CLINICAL TRIAL: NCT03831399
Title: Beneficial Effect of Leucine Supplementation in Muscular, Functional and Cognitive Functions in Sarcopenic Older Individuals
Brief Title: Leucine Supplementation in Sarcopenic Older Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Armonea Group - La Saleta (Unknown); Bonusan BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H1524420647893
Record Dates: First submitted 2018-11-09; First posted 2019-02-05 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2019-07

CONDITIONS: Frail Elderly Syndrome; Sarcopenia
Keywords: Frailty; Aged; Leucine; Sarcopenia
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — Leucine

STUDY DESIGN:
Intervention Model Description: Study of phase I, pilot, prospective, multicentric, randomized, double blind and placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Administration of Leucine or placebo (microcrystalline cellulose) will be done twice/day in the morning and in the afternoon for 13 weeks measuring spoon of placebo. Both products will be delivered in white jars, without label, and will carry the patient number on the outside. Randomization of numbers to either placebo or verum product will take place by Bonusan and will be revealed to the researchers at the end of final phase.
  The administration of prebiotics or placebo will last 13 weeks except for appearance of side-effects related to the study. The side-effects will be recorded and consulted with Bonusan Research Staff.
  The researcher enrolled in the geriatric, psychological or analytical measurements will be blind to the drug treatment.
  After finishing the study period, the study the Director of the Research group (Dr. Omar Cauli) will ask Bonusan to reveal who participants received Leucine and those who received placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Subjects in control group will receive placebo (lactose) 6g/day in two doses, in two spoon at noon (12 pm) and in the late afternoon (8 pm) for 13 weeks.
  The product will be delivered in powder, in white jars, without label, and will only carry the patient number on the outside, 4 jars per participant.
  Interventions: Dietary Supplement: Placebo
- Intervention Group (Active Comparator): Subjects in intervention group will receive leucine 6g/day, in tin two doses, in two spoon at noon (12 pm) and in the late afternoon (8 pm) for 13 weeks.
  The product will be delivered in powder, in white jars, without label, and will only carry the patient number on the outside, 4 jars per participant.
  Interventions: Dietary Supplement: Leucine

INTERVENTIONS:
Dietary Supplement: Leucine — Administration 6 g/day of leucine at noon (12 pm) and in the late afternoon (8 pm) for 13 weeks
  Arms: Intervention Group
Dietary Supplement: Placebo — Administration 6 g/day of lactose at noon (12 pm) and in the late afternoon (8 pm) for 13 weeks
  Arms: Control Group

SUMMARY:
Caring with older people in west societies has becoming a challenge for all health professional and any measure that can increase health or well-being will be ultimately improve quality of life and life expectancy. Frailty is a geriatric syndrome describing physical and functional decline that occurs as a consequence of certain diseases (e.g., cancer, chronic infection, etc.) but also even without disease. Frailty is characterized by an increased risk for poor outcomes such as incident falls, fractures, disability, comorbidity, health care expenditure and premature mortality. The aetiology of frailty is not well understood but it has been associated with changes in several physiologic systems, including inflammation, metabolic and micronutrients deficits.

The investigators wish to test with a confident perspective that any measured that improve the efficiency of muscular system can prevent the progression of frailty syndrome and that can have many others effects since it has been consistently demonstrated that a proper muscular function in aging is associated with other signs and symptoms. Looking at the literature, there are two clinical trials that evaluated the effect of leucine supplementation in older individuals with beneficial effects. The investigators wish to replicate those findings and to extend the analysis of the effect afforded by leucine supplementation in sarcopenia, frailty and cognitive function in individuals living in nursing homes in Valencia and province. This trial will show the eventual effects of leucine supplementation in elderly people may be also useful to afford some beneficial effects (sleep, cognitive function, depressed mood, balance and gait, etc) by modulating the function of muscular and metabolic system and in reduce the progression of sarcopenia and loss of muscular function.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk alone or with help of a can or a walker
* Age 60 years or older
* Cognitive function equal or higher than 21points in Mini-mental examination score
* Both genders
* Institutionalized in nursing homes for at least 6 months

Exclusion Criteria:

* Clinical diagnosed severe dementia
* Severe psychiatric disease (i.e. schizophrenia)
* Glomerular filtrate <30 ml/min/1,73m2

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Lean mass | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated according to European Group of Working Sarcopenia in older people criteria:
  Skeletal muscle mass index (kg/m2)
Strength | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated according to European Group of Working Sarcopenia in older people criteria:
  Handgrip Strength (kg)
Physical performance | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated according to European Group of Working Sarcopenia in older people criteria:
  Walking speed (m/s)

SECONDARY OUTCOMES:
Cholesterol | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated with a blood analysis to determine total, HDL and LDL cholesterol (mg/dL)
Glucose | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated with a blood analysis to determine glucose (mg/dL)
Creatinine | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated with a blood analysis to determine creatinine (mg/dL)
Triglycerides | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated with a blood analysis to determine triglycerides (mg/dL)
IL-6 | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as:
  IL6 (pg/mL)
TNF-alfa | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as:
  TNF-alfa (pg/mL)
IGF-1 | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as:
  IGF-1 (mg/mL)
Leucine | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as leucine concentration (mg/mL)
Valine | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as valine concentration (mg/mL)
Isoleucine | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as isoleucine concentration (mg/mL)
Glutamine | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as glutamine concentration (mg/mL)
B-alanine | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as B-alanine concentration (mg/mL)
Albumine | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as:
  albumine (g/L)
Transthyretin | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as:
  transthyretin (mg/L)
Myostatin | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, metabolic biomarkers related to sarcopenia and muscular function of all participants will be evaluated as:
  myostatin (ng/mL)
Body mass index | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated as:
  Body mass index (kg/m2)
Body perimeters | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated as:
  Abdominal and calf perimeter (cm)
Body composition | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated as bioimpedance to know fat and lean mass (kg)
Comorbidities | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated as Charlson index score (absence of comorbidity: 0-1 points, low comorbidity: 2 points, and high comorbidity > 3 points)
Type and number of drugs used | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, the drugs consumed by each participant will be collected
Gait and balance | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated with Tinetti index Scale(0 to 28 points, 19-24 risk of falling, <19 high risk of falling)
Basic activities of daily living | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated with Barthel index Scale to measure the activities of daily living and mobility (o to 100 points, < 60 dependence)
Cognitive performance | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated with Mini-mental score examination Scale (MMSE - 0 to 30 points, <24 points cognitive impairment, <21 mild cognitive impairment)
Depression | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated with Yesavage Scale for geriatric depression (0 to 15 points, >5 points high risk of depression)
Forced spirometry | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated as forced spirometry parameters (measured with a spirometer)
Respiratory muscles strenght | 4 months
  Before starting and after finishing administration of Leucine supplement or placebo, all participants will be evaluated as maximal respiratory pressures (measured with a respiratory pressure gauge)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Cauli, MD, PhD, Principal Investigator — Universitat de Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers

REFERENCES:
- [Derived] Buigues C, Theou O, Fonfria-Vivas R, Martinez-Arnau FM, Rockwood K, Cauli O. Can Leucine Supplementation Improve Frailty Index Scores? Geriatrics (Basel). 2023 Oct 12;8(5):102. doi: 10.3390/geriatrics8050102. PMID 37887975
- [Derived] Martinez-Arnau FM, Fonfria-Vivas R, Buigues C, Castillo Y, Molina P, Hoogland AJ, van Doesburg F, Pruimboom L, Fernandez-Garrido J, Cauli O. Effects of Leucine Administration in Sarcopenia: A Randomized and Placebo-controlled Clinical Trial. Nutrients. 2020 Mar 27;12(4):932. doi: 10.3390/nu12040932. PMID 32230954